CLINICAL TRIAL: NCT05457777
Title: The Effect of Motivational Interviews Based on Change Stages on the Digital Game Addiction Levels of Nursing Students
Brief Title: The Effect of Motivational Interviews on the Digital Game Addiction Levels of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidan Balkaya (Other)
Responsible Party: Sponsor-Investigator, Fidan Balkaya, Nursing-Master Student, Cumhuriyet University
Organization: Cumhuriyet University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sivas Cumhuriyet University
Record Dates: First submitted 2022-05-03; First posted 2022-07-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Motivational Interview; Addiction
Keywords: digital game addiction; nursing study; change stages; motivational interview
MeSH Terms: conditions — Behavior, Addictive | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Our study has two groups of 36 participants each. Our study is an experimental study with pretest-posttest control group.
Who Masked: Participant
Masking Description: Participants will be determined blindly by being assigned by a site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview group (Experimental): Motivational interviews will be held to the participants with digital game addiction in this group.
  Interventions: Behavioral: Motivational interview in digital game addiction
- Control group (No Intervention): This group will be control group and any motivational interviews will not be held to the participants with digital game addiction in this group.

INTERVENTIONS:
Behavioral: Motivational interview in digital game addiction — Motivational interviewing, which is a technique developed by William Miller that aims to change behavior by revealing the contradiction of problematic behavior with the value judgments of the person and creating motivation by the counselor, will be applied to the individuals with digital game addiction.
  Arms: Motivational interview group

SUMMARY:
The aim of this study is to reveal the effect of motivational interviewing based on change stages on digital game addiction. This study will be conducted with a total of 72 individuals assigned by a randomization site from all nursing students who study at Sivas Cumhuriyet University, Faculty of Health Sciences, voluntarily participated in the study, and were found to be digital game addicts. These individuals will be equally distributed to the intervention and control groups. Personal Information Form, Stages of Change Questionnaire and Digital Game Addiction Scale will be distributed to individuals to answer. The obtained data will be analyzed statistically.

DETAILED DESCRIPTION:
The aim of this study is to reveal the effect of motivational interviewing based on change stages on digital game addiction. This study will be conducted with a total of 72 individuals assigned by a randomization site from all nursing students who study at Sivas Cumhuriyet University, Faculty of Health Sciences, voluntarily participated in the study, and were found to be digital game addicts. These individuals will be equally distributed to the intervention and control groups. Each group will contain 36 participants. the participants in intervention group will take motivational interventions while the individuals who have digital game addiction in control group will not take this application. Personal Information Form, Stages of Change Questionnaire and Digital Game Addiction Scale will be distributed to individuals to answer. The obtained data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

Nursing students who:

* agree to participate in the study
* are over 18 years
* have game addiction
* agree to participate in the negotiations

Exclusion Criteria:

Individuals who:

* do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Digital Game Addiction Scale | up to three months
  The scale has a five-point Likert type, single-factor structure and scores between 1-5 (1=never, 5=always) (range: 7-35). Evaluation is made using monoetic and polyethical diagnoses. According to the monothetic diagnosis, if the person scores three (sometimes) or more on seven of the seven items; According to the polythetic diagnosis, if at least four of the seven items score three (sometimes) or more, it is defined as "game addict".

CONTACTS AND LOCATIONS:
Overall Officials: Semra Zorlu, PhD, Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers, they will be kept secret.